CLINICAL TRIAL: NCT05132010
Title: Prevalence of Gummy Smile: Cross-Sectional Study on A Sample of Egyptian Patients
Brief Title: Prevalence of Gummy Smile and Its Causes Among the Egyptian Population.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed mostafa ahmed abo el soud, resident at department of periodontology, Facult of Dentstry , Cairo university, Cairo University
Other Study IDs: prevalence of gummy smile
Record Dates: First submitted 2021-11-16; First posted 2021-11-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gummy Smile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
prevalence of gummy smile among the Egyptian population

DETAILED DESCRIPTION:
prevalence of gummy smile among Egyptian population in patients attending the kasr el aini hospital

ELIGIBILITY:
Inclusion Criteria:

* patients attending El kasr el Aini hospital at the department of periodontology.
* patients whose above 18 years old of both genders
* patients consulting the outpatient clinic
* provide informed consent

Exclusion Criteria:

* less than 18 years old
* patients having problems opening their mouth or undergoing inter maxillary fixation where oral examination will not be possible
* patients diagnosed with psychiatric problems or intoxicated with alcohol or drugs
* patients with gingival hyperplasia
* patients with extracted maxillary anterior teeth

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Egyptian population
Sampling Method: Non-Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
prevalence of gummy smile | through study completion, an average of 1 year
  To detect the prevalence of gummy smile among Egyptian population

SECONDARY OUTCOMES:
determining associated risk factors and classifying them onto further sub analytical groups | through study completion, an average of 1 year
  all the causes prevalence within the sample will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry , Cairo university, Giza, Egypt